CLINICAL TRIAL: NCT05595928
Title: Investigating Maternal Effects of Positions Applied in Patients Preparing for Caesarean Section Under Spinal Anesthesia
Acronym: cs position
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Aydin Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, ferdi gülaştı, Aydin Maternity and Child Health Hospital, Aydin Maternity and Child Health Hospital
Other Study IDs: 2022-10
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Patient Positioning

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Supine: supine
  Interventions: Other: position
- 15° left-lateral tilt position: 15° left-lateral tilt position.
  Interventions: Other: position
- 30° left-lateral tilt position.: 30° left-lateral tilt position.
  Interventions: Other: position

INTERVENTIONS:
Other: position — To compare whether there is a difference between maternal and fetal effects of Supine, 15-degree left tilt, and 30-degrees left tilt.

SUMMARY:
After the approval of the Ethics Committee, 120 patients were planned to be included in the study between 15.06.2022 and 15.01.2023. Women who underwent elective cesarean delivery under spinal anesthesia were randomized to the supine position, 15° left-lateral tilt position, or 30° left-lateral tilt position. The position will be changed to supine before the incision. It was planned to recruit 40 patients from each group, with a total of 120 patients. Anesthetic management was standardized and fluid administration with 10 mL/kg isotonic was planned. Hypotension (systolic blood pressure [SBP] reduction > 20% baseline or SBP <90 mm Hg) will be treated with intravenous bolus ephedrine based on maternal heart rate. The primary outcome is planned to include maternal SBP in 15 minutes of anesthesia induction, the amount of vasoactive drug administered before the end of surgery, and the incidence of hypotension during cesarean delivery.

DETAILED DESCRIPTION:
Pregnant women in the supine position may compress the Inferior Vena Cava (IVC) by compression of the enlarged uterus in the third trimester. In this way, it is considered that it may reduce the amount of returning blood and cause hypotension. The incidence of this condition, called Supine Hypotension Syndrome, was reported to be 8%-10% (1-3). Spinal anesthesia, decreased sympathetic tonus, decreased systemic vascular resistance, and vasodilation may also cause hypotension in the patient (4).

It was considered that if the uterus is tilted, the pressure on the IVC would be removed, increasing the return, blood volume and cardiac output, improving the fetus, blood supply and oxygen supply (5). However, studies that were conducted so far have not proven significant differences and there is no routine standard practice (6-8). Here, the purpose was to investigate the maternal effects between supine, tilt to the left of 15-degree, and tilt to the left of 30-degree., References

1. Howard BK, Goodson JH, Mengert WF. Supine hypotensive syndrome in late pregnancy. Obstet Gynecol. 1953;1:371-377.
2. Kinsella SM, Lohmann G. Supine hypotensive syndrome. Obstet Gynecol. 1994;83:774-788.
3. Rees GA, Willis BA. Resuscitation in late pregnancy. Anaesthesia. 1988;43:347-349.
4. Dyer RA, Reed AR, van Dyk D, et al. Hemodynamic effects of ephedrine, phenylephrine, and the coadministration of phenylephrine with oxytocin during spinal anesthesia for elective cesarean delivery. Anesthesiology. 2009;111:753-765.
5. Kinsella SM. Lateral tilt for pregnant women: why 15-degree? Anaesthesia. 2003;58:835-836.
6. Ellington C, Katz VL, Watson WJ, Spielman FJ. The effect of lateral tilt on maternal and fetal hemodynamic variables. Obstet Gynecol. 1991;77:201-203.
7. Bamber JH, Dresner M. Aortocaval compression in pregnancy: the effect of changing the degree and direction of lateral tilt on maternal cardiac output. Anesth Analg.

   2003;97:256-258.
8. Calvache JA, Mu.oz MF, Baron FJ. Hemodynamic effects of a right lumbar-pelvic wedge during spinal anesthesia for cesarean section. Int J Obstet Anesth. 2011;20:307-311.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery with term pregnancy
* Patient's height 150-180 cm
* American Society of Anesthesiologists (ASA) Physical Condition II
* Body Mass Index (BMI) <35 kg/m2.

Exclusion Criteria:

* Fetal macrosomia
* Uterine abnormalities (e.g. large fibroids, bicornuate uterus)
* Polyhydramnios
* Torn membranes, oligohydramnios
* Intrauterine growth restriction
* Gestational or non-gestational hypertension, diabetes, or eclampsia
* Contraindications for spinal anesthesia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since there are patients who will undergo cesarean section, female patients are included in the study.
Study Population: Women who underwent elective cesarean delivery under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-15 (Estimated); Study Completion 2023-01-15 (Estimated)

PRIMARY OUTCOMES:
position | through study completion, an average of 6 months
  the purpose was to investigate the maternal effects between supine, tilt to the left of 15-degree, and tilt to the left of 30-degree.

CONTACTS AND LOCATIONS:
Overall Officials: FERDİ GÜLAŞTI, Principal Investigator — Aydin Maternity and Child Health Hospital
Locations (1):
- Aydin Maternity and Child Health Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu T, Zou S, Guo L, Niu Z, Wang M, Xu C, Gao X, Shi Z, Guo X, Xiao H, Qi D. Effect of Different Positions During Surgical Preparation With Combined Spinal-Epidural Anesthesia for Elective Cesarean Delivery: A Randomized Controlled Trial. Anesth Analg. 2021 Nov 1;133(5):1235-1243. doi: 10.1213/ANE.0000000000005320. PMID 33350619